CLINICAL TRIAL: NCT06005259
Title: Effect of Spironolactone in the Prevention of Anthracycline-induced Cardiotoxicity: a Randomized Clinical Trial (SPIROTOX Trial)
Brief Title: Effect of Spironolactone in the Prevention of Anthracycline-induced Cardiotoxicity (SPIROTOX)
Acronym: SPIROTOX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar MD, PhD, Full Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SPIROTOX
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cardiotoxicity; Neoplasms; Chemotherapy Effect; Heart Failure
Keywords: Cardiotoxicity; Anthracyclines; Spironolactone
MeSH Terms: conditions — Cardiotoxicity; Neoplasms; Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will be administered 25 mg of spironolactone daily for 12 months, beginning 5 to 15 days prior to chemotherapy.
  Interventions: Drug: Spironolactone
- Control (Placebo Comparator): Participants will be given placebo daily for 12 months, beginning 5 to 15 days prior to chemotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Spironolactone 25 mg capsule
  Arms: Intervention
Drug: Placebo — Placebo capsule
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate the effect of spironolactone in the primary prevention of cardiotoxicity in cancer patients who are undergoing chemotherapy with anthracycline within 12 months. The main question it aims to answer is:

• Does spironolactone reduce the incidence of cardiotoxicity in patients undergoing anthracycline chemotherapy?

Participants will:

* Be cancer patients over 18 years starting treatment with anthracycline;
* Be randomized to receive either spironolactone or a placebo for 1 year;
* Undergo assessments of their left ventricular ejection fraction (LVEF), global longitudinal strain, and cardiac biomarkers over the 12-month period.

Researchers will compare the spironolactone group to the placebo group to see if cardiotoxicity incidence differs between the two.

DETAILED DESCRIPTION:
Objective:

To assess the potential of spironolactone in preventing anthracycline-induced cardiotoxicity among cancer patients.

Background:

There's ongoing debate and a dearth of evidence regarding the role of mineralocorticoid receptor antagonists, such as spironolactone, in averting anthracycline-induced cardiotoxicity.

Study Design:

A randomized, double-blind, placebo-controlled trial conducted at a single center.

Sample Size:

264 patients.

Intervention:

Eligible participants will be randomized on a 1:1 basis to either receive spironolactone or a placebo over a 12-month period.

Primary Outcome:

Incidence of cardiotoxicity at the 12-month mark.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer indicated for anthracycline chemotherapy treatment
* Age 18 and above
* Signed informed consent form

Exclusion Criteria:

* Previous use of anthracycline.
* Hypersensitivity to any mineralocorticoid receptor antagonists
* Symptoms of heart failure (exertional dyspnea, orthopnea, nocturnal paroxysmal dyspnea, and pulmonary or systemic congestion)
* Left ventricular ejection fraction (LVEF) < 45%
* Previous diagnosis of cardiomyopathy, coronary artery disease, or moderate to severe mitral or aortic disease
* Renal insufficiency defined as an estimated glomerular filtration rate < 30 ml/min/m2
* Hyperkalemia, defined as serum potassium ≥ 5.0 mmol/L
* Chronic liver disease, defined aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values more than 3 times the upper limit of normal
* Current participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity | 12 months
  Incidence of cardiotoxicity, defined as:
  * A decrease in ejection fraction (LVEF) by 10% or more to LVEF < 50%, as seen on transthoracic echocardiogram; OR
  * Relative drop in global longitudinal strain greater than 15% compared to baseline, observed on transthoracic echocardiogram; OR
  * New increase in cardiac biomarkers (troponin T > 99th percentile and/or NT-proBNP > 125 pg/mL).

SECONDARY OUTCOMES:
Left ventricular dysfunction | 3, 6 and 12 months
  Decrease in ejection fraction (LVEF) ≥ 10% to LVEF < 50% seen on transthoracic echocardiogram and cardiac magnetic resonance imaging
Ventricular function | 3, 6 and 12 months
  Relative reduction in global longitudinal strain ≥ 15%, observed on transthoracic echocardiogram and cardiac magnetic resonance imaging
Incidence of myocardial injury | 6 and 12 months
  Elevation of biomarkers (troponin T > 99th percentile and/or NT-proBNP > 125 pg/mL).
Oxygen consumption | 6 and 12 months
  Measurement of oxygen consumption (VO2), ventilatory equivalents for oxygen (VE/VO2) and for carbon dioxide (VE/VCO2) by cardiopulmonary exercise test
Ventricular diameters | 3, 6 and 12 months
  Ventricular diameters measured by transthoracic echocardiogram
Myocardial work | 3, 6 and 12 months
  Global work index (GWI) and global constructive work (GCW) measured by transthoracic echocardiogram
Diastolic dysfunction | 3, 6 and 12 months
  Assessment by echocardiography the incidence of diastolic dysfunction using the following parameters: peak E-wave velocity, peak A-wave velocity, mitral valve (MV) E/A ratio, MV deceleration time, pulsed-wave tissue doppler imaging e' velocity, Mitral E/e', left atrium maximum volume index, pulmonary vein(PV) systole(S) wave, PV diastole (D) wave, continuous wave (CW) doppler: tricuspid regurgitation, systolic jet velocity; Color M- mode.
Composite endpoint of mortality or major cardiovascular outcomes | 3, 6 and 12 months
  Composite endpoint of mortality or major cardiovascular outcomes (defined as acute myocardial infarction, symptomatic heart failure or complex arrhythmia).

OTHER OUTCOMES:
Quality of life measured by EQ-5D-3L (EuroQol 5 Dimension 3 Level) questionnaire | 3, 6 and 12 months
  The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, using 3 levels; 1 indicates better health state (no problems); 3 indicate worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Medication adherence | 3, 6 and 12 months
  Medication adherence rate measured by the Morisky-Green index
Oncological Treatment Discontinuation Rate | 12 months
Tumor Recurrence | 12 months
Hospitalization Rate | 12 months
Mortality Rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkatesh P, Kasi A. Anthracyclines. 2023 Jan 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538187/ PMID 30844214
- [Background] Barbosa RR, Bourguignon TB, Torres LD, Arruda LS, Jacques TM, Serpa RG, Calil OA, Barbosa LFM. Anthracycline-associated cardiotoxicity in adults: systematic review on the cardioprotective role of beta-blockers. Rev Assoc Med Bras (1992). 2018 Aug;64(8):745-754. doi: 10.1590/1806-9282.64.08.745. PMID 30673046
- [Background] Rawat PS, Jaiswal A, Khurana A, Bhatti JS, Navik U. Doxorubicin-induced cardiotoxicity: An update on the molecular mechanism and novel therapeutic strategies for effective management. Biomed Pharmacother. 2021 Jul;139:111708. doi: 10.1016/j.biopha.2021.111708. Epub 2021 May 13. PMID 34243633
- [Background] Cardinale D, Iacopo F, Cipolla CM. Cardiotoxicity of Anthracyclines. Front Cardiovasc Med. 2020 Mar 18;7:26. doi: 10.3389/fcvm.2020.00026. eCollection 2020. PMID 32258060
- [Background] Herrmann J, Lenihan D, Armenian S, Barac A, Blaes A, Cardinale D, Carver J, Dent S, Ky B, Lyon AR, Lopez-Fernandez T, Fradley MG, Ganatra S, Curigliano G, Mitchell JD, Minotti G, Lang NN, Liu JE, Neilan TG, Nohria A, O'Quinn R, Pusic I, Porter C, Reynolds KL, Ruddy KJ, Thavendiranathan P, Valent P. Defining cardiovascular toxicities of cancer therapies: an International Cardio-Oncology Society (IC-OS) consensus statement. Eur Heart J. 2022 Jan 31;43(4):280-299. doi: 10.1093/eurheartj/ehab674. PMID 34904661
- [Background] Kalay N, Basar E, Ozdogru I, Er O, Cetinkaya Y, Dogan A, Inanc T, Oguzhan A, Eryol NK, Topsakal R, Ergin A. Protective effects of carvedilol against anthracycline-induced cardiomyopathy. J Am Coll Cardiol. 2006 Dec 5;48(11):2258-62. doi: 10.1016/j.jacc.2006.07.052. Epub 2006 Nov 9. PMID 17161256
- [Background] Kaya MG, Ozkan M, Gunebakmaz O, Akkaya H, Kaya EG, Akpek M, Kalay N, Dikilitas M, Yarlioglues M, Karaca H, Berk V, Ardic I, Ergin A, Lam YY. Protective effects of nebivolol against anthracycline-induced cardiomyopathy: a randomized control study. Int J Cardiol. 2013 Sep 1;167(5):2306-10. doi: 10.1016/j.ijcard.2012.06.023. Epub 2012 Jun 22. PMID 22727976
- [Background] Avila MS, Ayub-Ferreira SM, de Barros Wanderley MR Jr, das Dores Cruz F, Goncalves Brandao SM, Rigaud VOC, Higuchi-Dos-Santos MH, Hajjar LA, Kalil Filho R, Hoff PM, Sahade M, Ferrari MSM, de Paula Costa RL, Mano MS, Bittencourt Viana Cruz CB, Abduch MC, Lofrano Alves MS, Guimaraes GV, Issa VS, Bittencourt MS, Bocchi EA. Carvedilol for Prevention of Chemotherapy-Related Cardiotoxicity: The CECCY Trial. J Am Coll Cardiol. 2018 May 22;71(20):2281-2290. doi: 10.1016/j.jacc.2018.02.049. Epub 2018 Mar 11. PMID 29540327
- [Background] Cardinale D, Colombo A, Sandri MT, Lamantia G, Colombo N, Civelli M, Martinelli G, Veglia F, Fiorentini C, Cipolla CM. Prevention of high-dose chemotherapy-induced cardiotoxicity in high-risk patients by angiotensin-converting enzyme inhibition. Circulation. 2006 Dec 5;114(23):2474-81. doi: 10.1161/CIRCULATIONAHA.106.635144. Epub 2006 Nov 13. PMID 17101852
- [Background] Livi L, Barletta G, Martella F, Saieva C, Desideri I, Bacci C, Del Bene MR, Airoldi M, Amoroso D, Coltelli L, Scotti V, Becherini C, Visani L, Salvestrini V, Mariotti M, Pedani F, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Olivotto I, Meattini I. Cardioprotective Strategy for Patients With Nonmetastatic Breast Cancer Who Are Receiving an Anthracycline-Based Chemotherapy: A Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1544-1549. doi: 10.1001/jamaoncol.2021.3395. PMID 34436523
- [Background] Omland T, Heck SL, Gulati G. The Role of Cardioprotection in Cancer Therapy Cardiotoxicity: JACC: CardioOncology State-of-the-Art Review. JACC CardioOncol. 2022 Mar 15;4(1):19-37. doi: 10.1016/j.jaccao.2022.01.101. eCollection 2022 Mar. PMID 35492815
- [Background] Wang Y, Lu X, Wang X, Qiu Q, Zhu P, Ma L, Ma X, Herrmann J, Lin X, Wang W, Xu X. atg7-Based Autophagy Activation Reverses Doxorubicin-Induced Cardiotoxicity. Circ Res. 2021 Oct;129(8):e166-e182. doi: 10.1161/CIRCRESAHA.121.319104. Epub 2021 Aug 13. PMID 34384247
- [Background] Akpek M, Ozdogru I, Sahin O, Inanc M, Dogan A, Yazici C, Berk V, Karaca H, Kalay N, Oguzhan A, Ergin A. Protective effects of spironolactone against anthracycline-induced cardiomyopathy. Eur J Heart Fail. 2015 Jan;17(1):81-9. doi: 10.1002/ejhf.196. Epub 2014 Nov 20. PMID 25410653
- [Background] Davis MK, Villa D, Tsang TSM, Starovoytov A, Gelmon K, Virani SA. Effect of Eplerenone on Diastolic Function in Women Receiving Anthracycline-Based Chemotherapy for Breast Cancer. JACC CardioOncol. 2019 Dec 17;1(2):295-298. doi: 10.1016/j.jaccao.2019.10.001. eCollection 2019 Dec. No abstract available. PMID 34396193
- [Background] Cardinale D, Colombo A, Bacchiani G, Tedeschi I, Meroni CA, Veglia F, Civelli M, Lamantia G, Colombo N, Curigliano G, Fiorentini C, Cipolla CM. Early detection of anthracycline cardiotoxicity and improvement with heart failure therapy. Circulation. 2015 Jun 2;131(22):1981-8. doi: 10.1161/CIRCULATIONAHA.114.013777. Epub 2015 May 6. PMID 25948538
- [Background] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Background] Laufer-Perl M, Perelman-Gvili M, Sirota Dorfman S, Baruch G, Rothschild E, Beer G, Arbel Y, Arnold JH, Rozenbaum Z, Banai S, Topilsky Y, Kapusta L. Prevalence of Right Ventricle Strain Changes following Anthracycline Therapy. Life (Basel). 2022 Feb 15;12(2):291. doi: 10.3390/life12020291. PMID 35207578